CLINICAL TRIAL: NCT03573414
Title: Gut Microbial Metabolism of Polyphenols and Cardiovascular Health
Brief Title: Gut Microbial Metabolism of Polyphenols and Cardiovascular Health (StratiPol) (Stratification Study)
Acronym: StratiPol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Washington Red Raspberry Commission (Other)
Responsible Party: Principal Investigator, Dr Ana Rodriguez-Mateos, Lecturer in Nutrition, King's College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Stratification Study
Record Dates: First submitted 2018-06-01; First posted 2018-06-29 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: Cardiovascular system; Polyphenols
MeSH Terms: interventions — Soy Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy men and women (Experimental): Intervention:
  2*breakfast containing 40 g of raspberry powder, 30 g milled flax seeds and 250 mL of soy Milk.
  Interventions: Other: raspberry powder, milled flaxseed and soy milk

INTERVENTIONS:
Other: raspberry powder, milled flaxseed and soy milk — * The participants will consume a breakfast consisting of 30 g of milled flaxseed, 40 g of raspberry powder and 250 ml of soy milk for 3 days
  * The participants will provide blood and urine samples

SUMMARY:
There is increasing interest in the effects of various food derived polyphenols on cardiovascular health. Several studies have demonstrated improvements in vascular function after intake of polyphenol rich foods. The objective of this study is to investigate the association between polyphenol microbiota metabolism and cardiovascular health.

The participants (n=250) with age range between 20 to 70 years old health overweight men and women. The participants will consume a polyphenol rich breakfast for three days (consisting on milled flaxseed, raspberry powder and soy milk). The participants will provide the investigators with urine and blood samples for polyphenol analysis. Cardiovascular measurements such as PWV, AIx, Blood Pressure and FMD will be performed at baseline and after 72h.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 20-70 years
* BMI between 18.5 and 35 kg/m2
* Subjects are willing to maintain their normal eating/drinking habits and exercise habits to avoid changes in body weight over the duration of the study
* Are able to understand the nature of the study
* Able to give signed written informed consent
* Signed informed consent form

Exclusion Criteria:

* Medical history of cardiovascular disease including coronary artery disease, cerebrovascular disease and peripheral artery disease
* Hypertensive, defined as 140/90mmHg or higher
* Obese participants with BMI superior or equal to 35 kg/m2
* Underweight participants defined by a BMI inferior to 18.5 kg/m2
* Medical history of diabetes mellitus, metabolic syndrome, terminal renal failure or malignancies
* Abnormal heart rhythm (lower or higher than 60-100 bpm)
* Allergies to berries or other significant food allergy
* Subjects under medication that can affect the cardiovascular system or on vitamin/dietary supplements.
* Subjects who have lost more than 10% of their weight in the past 6 months or are currently in a diet
* Subjects who reported participant in another study within one month before the study start
* Subjects who smoke an irregular amount of cigarettes per day
* Pregnant women or planning to become pregnant in the next 6 months
* Any reason or condition that in the judgment of the clinical investigator(s) may put the subject at unacceptable risk or that may preclude the subject from understanding or complying with the study's requirements.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Plasma and 24 h urine gut microbial polyphenol metabolites after high polyphenol breakfast. | 1-3 days
  To examine ellagitannins, lignans and isoflavones metabolites levels in urine and plasma assessed by liquid chromatography - mass spectrometer (LCMS) post 3 days consumption of high polyphenol breakfast contain 40 g raspberry powder, 30 g milled flaxseed and 250 mL soy milk to establish metabotypes.

SECONDARY OUTCOMES:
Changes in flow- mediated dilation after 3 days consumption of high polyphenol breakfast. | Baseline 0 and 72 hours.
  Determine the effect post 3 day consumption of a polyphenol rich breakfast containing raspberry ellagitannins, flaxseed lignans and soy milk isoflavones on endothelium-dependent flow mediated dilation (FMD) of the brachial artery, including diameter and flow velocity using Ultra sound device.
Changes in Pulse Wave Velocity (PWV) after 3 days consumption of high polyphenol. breakfast | Baseline 0 and 72 hours.
  Determine the effect post 3 days of consumption of a polyphenol rich breakfast containing raspberry ellagitannins, flaxseed lignans and soy milk isoflavones on arterial stiffness measured as pulse wave velocity (PWV) using a Sphygmocor device.
Changes in augmentation Index (AIx) after 3 days consumption of high polyphenol breakfast. | Baseline 0 and 72 hours.
  Determine the effect post 3 days of consumption of a polyphenol rich breakfast containing raspberry ellagitannins, flaxseed lignans and soy milk isoflavones on arterial stiffness measured Augmentation index ( AIX) using a Sphygmocor device.
Changes in office Blood pressure after 3 days consumption of high polyphenol breakfast. | Baseline 0 and 72 hours.
  Determine the effect post 3 days of consumption of a polyphenol rich breakfast containing raspberry ellagitannins, flaxseed lignans and soy milk isoflavones on central and peripheral systolic and diastolic blood pressure.
Changes in heart rate after 3 days consumption of high polyphenol breakfast. | Baseline 0 and 72 hours.
  Determine the effect post 3 days of consumption of a polyphenol rich breakfast containing raspberry ellagitannins, flaxseed lignans and soy milk isoflavones on heart rate.
Plasma and Urine polyphenol metabolites levels for ellagitannins, lignans and isoflavones. | Baseline 0 and 72 hours
  Determine the bioavailability of polyphenols post 3 days of consumption of a polyphenol rich breakfast in blood and urine samples measured by liquid chromatograph - mass spectrometry (LCMS)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ana Rodriguez-Mateos, PhD, Principal Investigator — ana.rodriguez-mateos@kcl.ac.uk
Locations (1):
- King's College London, Department of Nutritional Sciences, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No